CLINICAL TRIAL: NCT01727791
Title: A Multiple Dose Pharmacokinetic Open-label Study Of Pregabalin (Lyrica Registered) In Healthy Lactating Women
Brief Title: A Study Of Pregabalin (Lyrica) Drug Levels In Urine, Plasma And Breast Milk Of Healthy Lactating Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Other
Other Study IDs: A0081181; 2012-003197-57 (EudraCT Number)
Record Dates: First submitted 2012-11-12; First posted 2012-11-16 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2016-04

CONDITIONS: Healthy Lactating Women
Keywords: pharmacokinetic; pregabalin; lactation
MeSH Terms: conditions — Breast Feeding | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label (Experimental)
  Interventions: Drug: pregabalin (Lyrica)

INTERVENTIONS:
Drug: pregabalin (Lyrica) — Subjects will receive a single 150 mg dose of pregabalin in the evening of Day 1, a 150 mg dose of pregabalin in the morning and evening of Day 2 and a 150 mg dose in the morning of Day 3.

SUMMARY:
This is a pharmacokinetic study to determine the safety and tolerability of pregabalin in healthy lactating women. The objectives are to determine whether pregabalin is secreted in breast milk and if so, to characterize pregabalin pharmacokinetics in breast milk. Other objectives are to estimate potential infant exposure to pregabalin if administered to lactating women and to characterize the safety and tolerability of pregabalin in lactating women.

DETAILED DESCRIPTION:
Post approval commitment for the FDA

ELIGIBILITY:
Inclusion Criteria:

* Healthy lactating females between the ages of 18 and 45 years (inclusive) who are actively breast-feeding or expressing breast milk and are at least 12 weeks post partum.
* Subjects must be willing to temporarily discontinue breast feeding their infants before the Day 1 evening dose through to 42 hours after the last dose

Exclusion Criteria:

* History of significant adverse reaction to pregabalin or gabapentin.
* Subjects pregnant or unwilling or unable to comply with the Lifestyle guidelines presented in the protocol during the study period and through the follow-up visit.
* Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric (including post natal depression), neurologic or allergic disease (including drug allergies, but excluding untreated asymptomatic, seasonal allergies at time of dosing).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081181&StudyName=A%20Study%20Of%20Pregabalin%20%28Lyrica%29%20Drug%20Levels%20In%20Urine%2C%20Plasma%20And%20Breast%20Milk%20Of%20Healthy%20Lactating%20Women

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were healthy, lactating females between the ages of 18 and 45 years (inclusive) who were actively breastfeeding or expressing breast milk, who were at least 12 weeks post-partum and not currently pregnant.
Groups:
- Pregabalin: Participants received pregabalin 150 milligram (mg) immediate-release (IR) capsule over 12-hour dosing intervals on Day 1, Day 2 and Day 3.
Period: Overall Study
Arm/Group | Pregabalin
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included participants who received at least 1 dose of study medication.
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau)
Description: Area under the plasma concentration-time profile from time 0 to tau (AUCtau), where tau was the dosing interval of 12 hours.
Time Frame: Pre-dose on Day 3; 0.5, 1, 2, 3, 4, 6, 10, 12 hours post-dose on Day 3
Population: The pharmacokinetic (PK) parameter analysis population included participants who received study medication and who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter (mcg*hr/mL)
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
microgram*hour/milliliter (mcg*hr/mL) | 32.50 (24)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax was the peak concentration in plasma post Day 3 dose.
Time Frame: Pre-dose on Day 3; 0.5, 1, 2, 3, 4, 6, 10, 12, 18, 24 hours post-dose on Day 3
Population: The PK parameter analysis population included participants who received study medication and who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
mcg/mL | 4.67 (18)

3. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: Tmax was the time to peak concentration in plasma post Day 3 dose.
Time Frame: Pre-dose on Day 3; 0.5, 1, 2, 3, 4, 6, 10, 12, 18, 24 hours post-dose on Day 3
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
hr | 2.01 [1.00 to 3.00]

4. Primary Outcome: Plasma Half-Life (t1/2)
Description: Plasma decay half-life (t1/2) was the time for the plasma concentration to decrease by one-half. The t1/2 is based on the terminal elimination phase time points from this timeframe.
Time Frame: Pre-dose on Day 3; 0.5, 1, 2, 3, 4, 6, 10, 12, 18, 24 hours post-dose on Day 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
hr | 5.624 (0.65656)

5. Primary Outcome: Average Plasma Concentration During the Dosing Interval (Cav)
Description: Average plasma concentration during the dosing interval (Cav) was calculated by dividing AUCtau (plasma) with tau, where tau was the dosing interval of 12 hours.
Time Frame: Pre-dose on Day 3; 0.5, 1, 2, 3, 4, 6, 10, 12 hours post-dose on Day 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
mcg/mL | 2.709 (24)

6. Primary Outcome: Minimum Observed Plasma Trough Concentration (Cmin)
Description: Cmin was the minimum observed plasma concentration of a drug after post Day 3 dose.
Time Frame: Pre-dose on Day 3; 0.5, 1, 2, 3, 4, 6, 10, 12, 18, 24 hours post-dose on Day 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
mcg/mL | 1.246 (36)

7. Primary Outcome: Apparent Oral Clearance (CL/F)
Description: Apparent oral clearance (CL/F) was calculated by dividing dose by the AUCtau, where tau was the dosing interval of 12 hours. Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Pre-dose on Day 3; 0.5, 1, 2, 3, 4, 6, 10, 12 hours post-dose on Day 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/minute
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
mL/minute | 76.90 (24)

8. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval for Breast Milk (AUCtau [Breast Milk])
Description: AUCtau (breast milk) was the area under the curve for breast milk, from time 0 to tau (AUCtau), where tau was the dosing interval of 12 hours.
Time Frame: Pre-dose on Day 3; 0 to 2, 2 to 4, 4 to 8, 8 to 12 hours post-dose on Day 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
mcg*hr/mL | 24.64 (27)

9. Primary Outcome: Maximum Observed Concentration in Breast Milk (Cmax [Breast Milk])
Description: Cmax (breast milk) was the maximum observed concentration in breast milk post Day 3 dose.
Time Frame: Pre-dose on Day 3; 0 to 2, 2 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 32, 32 to 40 and 40 to 48 hours post-dose on Day 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
mcg/mL | 2.474 (30)

10. Primary Outcome: Time to Reach Maximum Observed Breast Milk Concentration (Tmax [Breast Milk])
Description: Tmax (breast milk) was time of the maximum observed breast milk concentration Day 3 post-dose.
Time Frame: Pre-dose on Day 3; 0 to 2, 2 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 32, 32 to 40 and 40 to 48 hours post-dose on Day 3
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
hr | 4.63 [3.08 to 6.16]

11. Primary Outcome: Terminal Half-Life for Breast Milk (t1/2 [Breast Milk])
Description: The terminal half-life for breast milk (t1/2 [breast milk]) was the time measured for breast milk concentration to decrease by one-half. For the first 5 participants enrolled under protocol amendment dated: 18 Sep 2012, breast milk was collected up to 24 hours after Day 3 dosing over the following time intervals: 0 to 2, 2 to 4, 4 to 8, 8 to 12, 12 to 24 hours. Terminal half-life was determined over those points characterizing the elimination phase. For the remaining 5 participants, there were 3 additional collection intervals (24 to 32, 32 to 40, 40 to 48 hours) for characterizing the terminal elimination phase. The t1/2 (breast milk) is based on the terminal elimination phase time points from this timeframe.
Time Frame: Pre-dose on Day 3; 0 to 2, 2 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 32, 32 to 40 and 40 to 48 hours post-dose on Day 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
hr | 8.117 (3.0871)

12. Primary Outcome: Average Breast Milk Concentration During the Dosing Interval (Cav)
Description: Average breast milk concentration during the dosing interval (Cav) was calculated by dividing AUCtau (breast milk) with tau, where tau was the dosing interval of 12 hours.
Time Frame: Pre-dose on Day 3; 0 to 2, 2 to 4, 4 to 8, 8 to 12 hours post-dose on Day 3
Population: as for outcome 2
Measure: Mean (Full Range); unit: mcg/mL
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
mcg/mL | 2.116 (27) [1.34 to 3.06]

13. Primary Outcome: Amount Excreted in Breast Milk Over the Dosing Interval Tau (Aetaubm)
Description: Aetaubm was the amount excreted in breast milk over the dosing interval tau (12 hours). It was calculated as the sum of (breast milk concentration * sample volume) for each collection interval from 0 to 12 hours post-dose, where tau was the dosing interval of 12 hours. Sample volume was based on ratio of volume weight and density.
Time Frame: Pre-dose on Day 3; 0 to 2, 2 to 4, 4 to 8, 8 to 12 hours post-dose on Day 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
mcg | 286.9 (60)

14. Primary Outcome: Percentage of Dose Excreted in Breast Milk During the Dosing Interval Tau (Aetaubm Percent)
Description: Percentage of dose excreted in breast milk during the dosing interval tau (Aetaubm percent) was calculated by using the formula: 100*(Aetaubm [sum of {breast milk concentration * sample volume} for each collection interval from 0 to 12 hours post-dose] divided by dose), where tau was the dosing interval of 12 hours.
Time Frame: Pre-dose on Day 3; 0 to 2, 2 to 4, 4 to 8, 8 to 12 hours post-dose on Day 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
percentage of dose | 0.1913 (60)

15. Primary Outcome: Breast Milk Clearance (CLbm)
Description: Breast milk clearance (CLbm) was calculated by dividing Aetaubm (sum of [breast milk concentration * sample volume] for each collection interval from 0 to 12 hours post-dose) by plasma AUCtau, where tau was the dosing interval of 12 hours.
Time Frame: Plasma: Pre-dose on Day 3; 0.5, 1, 2, 3, 4, 6, 10, 12 hours post-dose on Day 3. Breast milk: Pre-dose on Day 3; 0 to 2, 2 to 4, 4 to 8, 8 to 12 hours post-dose on Day 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
mL/min | 0.1473 (60)

16. Primary Outcome: Amount Recovered in Urine During the Dosing Interval Tau (Aetauurine)
Description: Aetauurine was the amount excreted in urine over the dosing interval tau (12 hours). It was calculated as the sum of (urine concentration * sample volume) for each collection interval from 0 to 12 hours post-dose, where tau was the dosing interval of 12 hours. Here, sample volume was based on the ratio of volume weight and density.
Time Frame: Pre-dose on Day 3; 0 to 2, 2 to 4, 4 to 8, 8 to 12 hours post-dose on Day 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
mg | 133.1 (12)

17. Primary Outcome: Percent of Dose Recovered in Urine During the Dosing Interval Tau (Aetauurine Percent)
Description: Percent of dose recovered in urine during the dosing interval tau (Aetauurine percent) was calculated as 100* (Aetau [sum of {urine concentration * sample volume} for each collection interval from 0 to 12 hours post-dose] divided by the dose), where tau was the dosing interval of 12 hours.
Time Frame: Pre-dose on Day 3; 0 to 2, 2 to 4, 4 to 8, 8 to 12 hours post-dose on Day 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
percentage of dose | 88.6 (12)

18. Primary Outcome: Renal Clearance (CLr)
Description: Renal clearance (CLr) was the volume of plasma from which the drug was completely removed by the kidney in a given amount of time. It was calculated by dividing Aetauurine (sum of [urine concentration * sample volume] for each collection interval from 0 to 12 hours post-dose) with the plasma AUCtau, where tau was the dosing interval of 12 hours.
Time Frame: Plasma: Pre-dose on Day 3; 0.5, 1, 2, 3, 4, 6, 10, 12 hours post-dose on Day 3. Urine: Pre-dose on Day 3; 0 to 2, 2 to 4, 4 to 8 and 8 to 12 hours post-dose on Day 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
mL/min | 68.16 (24)

19. Primary Outcome: Daily Amount of Pregabalin Excreted in Breast Milk (Ae24bm)
Description: Ae24bm was the daily amount of pregabalin excreted in breast milk. It was calculated by the formula: 2 * Aetaubm (sum of [breast milk concentration * sample volume] for each collection interval from 0 to 12 hours post-dose), where tau was the dosing interval of 12 hours.
Time Frame: Pre-dose on Day 3; 0 to 2, 2 to 4, 4 to 8, 8 to 12 hours post-dose on Day 3
Population: as for outcome 2
Measure: Mean (Full Range); unit: mcg
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
mcg | 664.6 (60) [270 to 1720]

20. Primary Outcome: Milk to Plasma Ratio for AUCtau (MPAUCtau)
Description: MPAUCtau was the ratio of AUCtau (breast milk) to AUCtau (plasma), where tau was the dosing interval of 12 hours.
Time Frame: as for outcome 15
Population: as for outcome 2
Measure: Mean (Full Range); unit: ratio
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
ratio | 0.769 [0.493 to 0.956]

21. Primary Outcome: Milk to Plasma Ratio for Maximum Observed Concentration (MPCmax)
Description: Milk to plasma ratio for maximum observed concentration (MPCmax) was calculated as the ratio of Cmax (breast milk) to Cmax (plasma).
Time Frame: Plasma: Pre-dose on Day 3; 0.5, 1, 2, 3, 4, 6, 10, 12, 18, 24 hours post-dose on Day 3. Breast milk: Pre-dose on Day 3; 0 to 2, 2 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 32, 32 to 40 and 40 to 48 hours post-dose on Day 3
Population: as for outcome 2
Measure: Mean (Full Range); unit: ratio
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
ratio | 0.5413 [0.335 to 0.755]

22. Primary Outcome: Body Weight Normalized Infant Dose (BWNID)
Description: Body weight normalized infant dose (BWNID) of pregabalin was the dose that an infant received from breast-feeding and was calculated from the milk to plasma AUCtau ratio multiplied by the average maternal plasma pregabalin concentration (Cav) multiplied by the standardized milk consumption for an infant (150 milliliter/kilogram/day [mL/kg/day]), where tau was the dosing interval of 12 hours.
Time Frame: as for outcome 15
Population: as for outcome 2
Measure: Mean (Full Range); unit: mcg/kg/day
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
mcg/kg/day | 317.3 (27) [202 to 458]

23. Primary Outcome: Body Weight Normalized Maternal Dose (BWNMD)
Description: Body weight normalized maternal dose (BWNMD) was calculated as the maternal dose in microgram per day (mcg/day) divided by maternal weight in kilogram (kg) at screening.
Time Frame: Pre-dose to 24 hours post-dose on Day 3
Population: as for outcome 2
Measure: Mean (Full Range); unit: mcg/kg/day
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
mcg/kg/day | 4343.6 (27) [3444 to 5676]

24. Primary Outcome: Infant Dose Expressed as Percentage of Body Weight Normalized Maternal Dose (BWNIDPCM)
Description: Infant dose expressed as percentage of body weight normalized maternal dose (BWNIDPCM) was the relative infant dose (relative to maternal dose) calculated by the formula: 100 * BWNID (Body Weight Normalized Infant Dose) / Body Weight Normalized Maternal Dose (BWNMD), where tau was the dosing interval of 12 hours.
Time Frame: Pre-dose to 24 hours post-dose on Day 3
Population: as for outcome 2
Measure: Mean (Full Range); unit: percentage of dose
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
percentage of dose | 7.341 (27) [4.43 to 9.78]

25. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to 28 days after last dose of study drug
Population: The safety analysis population included participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
participants
  Number of Participants with AEs | 8
  Number of Participants with SAEs | 0

26. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities
Description: The following parameters were analyzed for laboratory abnormalities: hematology (hemoglobin, hematocrit, red blood cell count, mean corpuscular volume [MCV], mean corpuscular hemoglobin [MCH], mean corpuscular hemoglobin concentration [MCHC], platelets, white blood cell count, lymphocytes, total neutrophils, basophils, eosinophils, monocytes); liver function (bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, total protein, albumin); renal function (blood urea nitrogen, creatinine, uric acid); electrolytes (sodium, potassium, chloride, calcium, bicarbonate); clinical chemistry (glucose); urinalysis (urine pH, glucose, ketones, protein, urine blood/hemoglobin, nitrite).
Time Frame: Baseline up to 28 days after last dose of study drug
Population: The safety analysis population included participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
participants | 4

27. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: The following parameters were analyzed for examination of vital signs: electrocardiogram (ECG), systolic and diastolic blood pressure, temperature, pulse rate, respiratory rate, radial pulse and body temperature.
Time Frame: Baseline up to 28 days after last dose of study drug
Population: The safety analysis population included participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 10
participants | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study drug
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=10)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 6 (9)
Headache (Nervous system disorders) | 2 (2)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.